CLINICAL TRIAL: NCT01116778
Title: A Phase III, Double-blind, Randomized, Parallel, Placebo-controlled Study to Evaluate the Efficacy and Safety of Probiotics eN-Lac® Capsules (Lactobacillus Paracasei GMNL-32) for the Treatment of Children With Perennial Allergic Rhinitis
Brief Title: the Efficacy and Safety of Probiotics eN-Lac® Capsules of Children With Perennial Allergic Rhinitis
Acronym: PAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GenMont Biotech Incorporation (Industry)
Collaborators: Biomedical Development Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MA0809005101
Record Dates: First submitted 2010-04-30; First posted 2010-05-05 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-08

CONDITIONS: Perennial Allergic Rhinitis; Probiotics; Lactobacillus Paracasei GMNL-32 (eN-Lac®)
Keywords: perennial allergic rhinitis; probiotics; Lactobacillus paracasei GMNL-32 (eN-Lac®); efficacy and safety
MeSH Terms: conditions — Rhinitis, Allergic, Perennial

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- eN-Lac® Capsules (Experimental)
  Interventions: Biological: eN-Lac®
- Placebo Capsules (Other)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: eN-Lac® — One capsule with 2x10^9 colony forming unit (cfu) LP GMNL-32, once daily, po
  Other Names: eN-Lac® Capsules (Lactobacillus paracasei GMNL-32)
  Arms: eN-Lac® Capsules
Other: Placebo — One placebo capsule, once daily, po
  Other Names: Placebo Capsules
  Arms: Placebo Capsules

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of probiotics eN-Lac® capsules (Lactobacillus paracasei GMNL-32) for the treatment of children with perennial allergic rhinitis(PAR).

DETAILED DESCRIPTION:
This study is PhaseIII clinical trial. According the results of PhaseII study,we find out the optimal dose and its maximum effectiveness in relieving the nasal symptoms of eN-Lac® (Lactobacillus paracasei GMNL-32) in children with PAR.

ELIGIBILITY:
Inclusion Criteria

* Subjects in age of 5-16 years old
* Subjects with a history of perennial allergic rhinitis for at least 1 year.
* Subjects with anyone of the following allergy test results (test results within 12 months before study are acceptable)
* Skin-Prick test:

Wheal diameter 3 mm larger than the negative control (salt water) and at least 1/2 the diameter of the positive control (histamine)

* Positive reaction determined by the CAP system Positive reaction defined as CAP score≥2
* Positive reaction determined by the MAST system Positive reaction defined as MAST score≥1
* Subject's mean nasal total symptom score (NTSS) throughout the screening period (4 to 10 days) should be ≥ 5 and ≤ 10; at least 3 days should be recorded during the screening period
* Subjects' parents or their legally acceptable representatives have signed the informed consent form.

Exclusion Criteria

* Subjects have clinically significant laboratory abnormality results (hematology, biochemistry or urinalysis tests) as determined by the investigator (tests performed during 14 days prior to visit 1 or during baseline period can be used for evaluating those criteria).
* Subjects with acute or significant chronic sinusitis, severe persistent asthma, congenital immunodeficiency, massive wound in oral cavity, use of rhinitis medications, neuropsychiatric disorders, immunocompromised, or chronic use of tricyclic antidepressants.
* Subjects need to take prohibited medications during the study or take the medications within the corresponding time frame indicated prior to the screening visit:

Parenteral or oral corticosteroids 30 days Nasal corticosteroids 30 days Topical use of flurandrenolide 30 days Topical use of clobetasol propionate 30 days Topical use of halobetasol propionate 30 days Astemizole 30 days Ketotifene 21 days Nedocromil or Sodium cromoglycate 14 days Loratadine 10 days Cetirizine 7 days Antileukotrienes 7 days Other H1 antihistamine 3 days Nasal decongestant 3 days Any food supplements including probiotics 3 days

* Subjects are undergoing desensitization therapy within 3 months prior to the screening period or subjects with vasomotor rhinitis.
* Subjects have participated investigational drug trial within 4 weeks before entering this study.
* Subjects are pregnant, lactating or planning to become pregnant.
* Subjects with any other serious diseases considered by the investigator that could interfere with the performance of NTSS result.
* Women of childbearing potential who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period.
* Subjects who is lack of physical integrity of gastrointestinal tract, or malabsorption syndrome, or inability to take oral medication.

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 236 (Actual)
Dates: Start 2010-05; Primary Completion 2012-01 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy profile of probiotics Lactobacillus paracasei GMNL-32 (eN-Lac®) in children with perennial allergic rhinitis. | NTSS is recorded daily on subject's DRC (daily record card) at the 8th week from baseline.
  NTSS is determined by the severity of allergic symptoms, including sneezing, rhinorrhea, nasal itching, and nasal stuffiness. These symptoms are evaluated using a four-point scale, namely, 0 = Absent, 1 = Mild (present but not disturbing), 2 = Moderate (disturbing but not hampering daytime activities and/or sleep), 3 = Severe (hampering daytime activities and/or sleep). NTSS is calculated by the sum of the scores of the symptoms.

SECONDARY OUTCOMES:
The safety features are evaluated through the changes of vital signs, physical examinations, laboratory test result (hematology, biochemistry and urinalysis tests), as well as the occurrence of adverse event. | at 8th week from basline
  The incidence of adverse events will be categorized by severity and related to the time of occurrence. Changes in physical examinations, changes in laboratory test results (hematology, biochemistry and urinalysis tests) from screening period, and change of vital signs will be summarized and analyzed by the descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Ying-Chen Lu, PhD, Study Director — GenMont Biothech Incorporation
Locations (4):
- Taiwan (4):
  - Taipei City Hospital Renai Branch, Taipei, Taipei
  - MacKay Memorial Hospital, Taipei, Taipei
  - Chang Gung Children's Hospital, Taipei, Taipei
  - Cardinal Tien Hospital, Xindian, Taipei